CLINICAL TRIAL: NCT03879980
Title: Effect of Preincisional Ultrasound-guided Quadratus Lumborum Block on Perioperative Analgesia and Inflammatory Responses in Transperitoneal Laparoscopic Nephrectomy: A Single-Blinded, Randomised Control Trial
Brief Title: Effect of Quadratus Lumborum Block on Perioperative Analgesia and Inflammatory Responses in Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Principal Investigator, Head of Intensive Care Unit, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes031
Record Dates: First submitted 2019-03-12; First posted 2019-03-19 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Pain
Keywords: quadratus lumborum block; pre-emptive analgesia; laparoscopic nephrectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Forty-four healthy patients with American Society of Anesthesiologists (ASA) classification I or II gave written consent to participate and were randomly allocated into QL block group or control (non-QL block) group. Randomisation used blocks of 4 into 2 groups using a list of random numbers and was performed by sealed envelopes. The surgeries were performed by 3 urology surgeon consultants with comparable distributions. Patients and principal investigator were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-QL block (Placebo Comparator): The control (non-QL block) group only received fentanyl IV during surgery.
  Interventions: Drug: Non-QL block
- Bilateral QL block (Experimental): The patients were in the semi-lateral supine position to show up the side to be blocked. Using USG and 1-6 MHz convex transducer placed in the transverse plane above the iliac crest at the level of the umbilicus. A Stimuplex® 20G 100-mm needle was advanced in anteroposterior direction toward the junction of tapered abdominal muscle layer and QL muscle, and 20 ml of 0.25% bupivacaine was deposited in the anterolateral border of QL muscle at the junction with the transversalis fascia reach outside the anterior layer of transversalis fascia. The lateral approach QL (type I) blocks were performed at both sides of patients. The total amount of bupivacaine was 100 mg for each patient
  Interventions: Drug: Bilateral QL block

INTERVENTIONS:
Drug: Bilateral QL block — Bilateral lateral Quadratus Lumborum block using 20 ml of 0.25% bupivacaine each injection as preemptive analgesia.
  Arms: Bilateral QL block
Drug: Non-QL block — Only received fentanyl IV during surgery.
  Arms: Non-QL block

SUMMARY:
Quadratus lumborum (QL) block can reduce intraoperative opioid consumption, decrease inflammation responses of IL-6, and reduce acute pain intensity in comparison with non-receiving QL block as the control group.

DETAILED DESCRIPTION:
Quadratus lumborum block had been studied as an effective postoperative analgesia in lower abdominal surgery, due to its spread to the thoracic paravertebral space and thoracolumbar fascia nerve. The effect of preincisional ultrasound (US)-guided QL block as "preemptive analgesia" on patient underwent laparoscopic living donor nephrectomy has never been evaluated. As preemptive analgesia, quadratus lumborum block could provide analgesics before and after surgery. Both groups immediately received basic postoperative analgesia regimen paracetamol 1 gr IV 8th hourly.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30 kg/m2
* ASA 1 or 2

Exclusion Criteria:

* refused to participate
* chronic use of analgesics or anti-inflammatory drugs
* allergy to local anaesthetic
* duration of surgery <4 or > 6 hours
* duration of anaesthesia <5 or > 7 hours
* neuropathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperative
  Intraoperative fentanyl consumption was recorded as total consumption in µg, and calculated into mean consumption per hour in µg.kg-1.h-1, due to the influence of patients body weight and duration of surgery to the given dose of fentanyl boluses.
Changes in Interleukin-6 from baseline | 24 hours
  Measurement of plasma Interleukin-6 before the anaesthesia induction as the baseline; 2 hours of surgical stimulation and gas insufflation intraoperatively; and 2 hours after recovery from anaesthesia.

SECONDARY OUTCOMES:
Numerical Rating Scale | 24 hours
  Pain measurement using Numerical Rating Scale (NRS) at rest and during movement. NRS from 0 =no pain to 10= worst pain at 2 hours and 24 hours after anaesthesia recovery
Hemodynamic Profiles: Heart Rate in bpm | Intraoperative
  The trends of perioperative haemodynamic profiles during and after surgery: heart rate in beat per minute
Hemodynamic Profiles: Systolic, Diastolic, and Mean Arterial Pressure in mmHg | Intraoperative
  The trends of perioperative haemodynamic profiles during and after surgery : systolic, diastolic and mean arterial pressure in mmHg
Number of participants with additional intravenous tramadol | 24 hours
  During observation after surgery, when the NRS began to increase > 3 at rest the intermittent tramadol 50 mg IV boluses was given 8th hourly. If the NRS still remained > 3, the intermittent tramadol 50 mg IV boluses were administered more frequently up to 4th hourly.
Number of participants with additional intravenous fentanyl | 24 hours
  If the pain relief was still inadequate after increasing tramadol boluses, the extra fentanyl 1 µg.kg^-1 IV boluses was given at every 15-30th minute until the NRS ≤ 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Hayden P, Cowman S. Anaesthesia for laparoscopic surgery. Continuing Education in Anaesthesia, Critical Care & Pain 2011;11(5):177-80.
- [Background] Barreveld A, Witte J, Chahal H, Durieux ME, Strichartz G. Preventive analgesia by local anesthetics: the reduction of postoperative pain by peripheral nerve blocks and intravenous drugs. Anesth Analg. 2013 May;116(5):1141-1161. doi: 10.1213/ANE.0b013e318277a270. Epub 2013 Feb 13. PMID 23408672
- [Background] Richebe P, Rivat C, Liu SS. Perioperative or postoperative nerve block for preventive analgesia: should we care about the timing of our regional anesthesia? Anesth Analg. 2013 May;116(5):969-970. doi: 10.1213/ANE.0b013e31828843c9. No abstract available. PMID 23606468
- [Background] Meleine M, Rivat C, Laboureyras E, Cahana A, Richebe P. Sciatic nerve block fails in preventing the development of late stress-induced hyperalgesia when high-dose fentanyl is administered perioperatively in rats. Reg Anesth Pain Med. 2012 Jul-Aug;37(4):448-54. doi: 10.1097/AAP.0b013e318257a87a. PMID 22660486
- [Background] de Oliveira CM, Sakata RK, Issy AM, Gerola LR, Salomao R. Cytokines and pain. Rev Bras Anestesiol. 2011 Mar-Apr;61(2):255-9, 260-5, 137-42. doi: 10.1016/S0034-7094(11)70029-0. English, Portuguese, Spanish. PMID 21474032
- [Background] Vadivelu N, Mitra S, Schermer E, Kodumudi V, Kaye AD, Urman RD. Preventive analgesia for postoperative pain control: a broader concept. Local Reg Anesth. 2014 May 29;7:17-22. doi: 10.2147/LRA.S62160. eCollection 2014. PMID 24872720
- [Background] Krohg A, Ullensvang K, Rosseland LA, Langesaeter E, Sauter AR. The Analgesic Effect of Ultrasound-Guided Quadratus Lumborum Block After Cesarean Delivery: A Randomized Clinical Trial. Anesth Analg. 2018 Feb;126(2):559-565. doi: 10.1213/ANE.0000000000002648. PMID 29135590
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] Warle MC, Berkers AW, Langenhuijsen JF, van der Jagt MF, Dooper PM, Kloke HJ, Pilzecker D, Renes SH, Wever KE, Hoitsma AJ, van der Vliet JA, D'Ancona FC. Low-pressure pneumoperitoneum during laparoscopic donor nephrectomy to optimize live donors' comfort. Clin Transplant. 2013 Jul-Aug;27(4):E478-83. doi: 10.1111/ctr.12143. Epub 2013 Jun 24. PMID 23795745
- [Background] Agarwal A, Yadav G, Gupta D, Singh PK, Singh U. Evaluation of intra-operative tramadol for prevention of catheter-related bladder discomfort: a prospective, randomized, double-blind study. Br J Anaesth. 2008 Oct;101(4):506-10. doi: 10.1093/bja/aen217. Epub 2008 Jul 24. PMID 18653496
- [Background] Moeller-Bertram T, Ky L, Coe C, Strigo I, Kincaid M, Keltner J, et al. Correlation of pain ratings and systemic interleukin-6 release in response to intramuscular capsaicin in healthy Humans. J Pain 2012;13(4):S52.
- [Background] Blanco R. TAP block under ultrasound guidance: the description of a "no pops" technique [Abstract]. Reg Anesth Pain Med 2007;32:S1-S130.
- [Background] Jianda X, Yuxing Q, Yi G, Hong Z, Libo P, Jianning Z. Impact of Preemptive Analgesia on inflammatory responses and Rehabilitation after Primary Total Knee Arthroplasty: A Controlled Clinical Study. Sci Rep. 2016 Aug 31;6:30354. doi: 10.1038/srep30354. PMID 27578313
- [Background] Farouk S. Pre-incisional epidural magnesium provides pre-emptive and preventive analgesia in patients undergoing abdominal hysterectomy. Br J Anaesth. 2008 Nov;101(5):694-9. doi: 10.1093/bja/aen274. Epub 2008 Sep 26. PMID 18820247